CLINICAL TRIAL: NCT06359951
Title: Implementation of Digital Brief, Scalable Single Session Interventions in Specialty Adolescent Care
Brief Title: Implementation of Project YES in Ambulatory Adolescent & Young Adult Medicine
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: American Psychological Association Division 53 Society for Clinical Child & Adolescent Psychology (Unknown)
Responsible Party: Principal Investigator, Anna Ros, Assistant Professor, Adolescent and Young Adult Psychologist, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0103
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Depression; Eating Disorders; Anxiety
MeSH Terms: conditions — Depression; Feeding and Eating Disorders; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Project YES (Experimental): This is a digital, self-guided SSI that has 3 options, Project Personality, Project CARE, and the ABC project. These teach adolescents about CBT skills including growth mindset, neutral self-talk and behavioral activation. Each option contains self-reflection exercises, vignettes from fictional peers, and psychoeducation that support users in understanding each CBT skill.
  See all materials for this intervention here: https://www.schleiderlab.org/yes.html
  Interventions: Behavioral: Project YES

INTERVENTIONS:
Behavioral: Project YES — Digital SSI

SUMMARY:
This study tests a suite of single-session intervention (SSI) targeting risk factors for depression and eating disorders among adolescents and young adults. Youth ages 13-25 who screen positive for depression or anxiety as a part of routine care will be offered one of three digital SSIs. Participants will complete questionnaires before the intervention, immediately after the intervention, and 3-months after completing the intervention so that the study team can investigate if Project YES leads to reductions in depression, anxiety and eating disorder symptoms.

ELIGIBILITY:
Inclusion Criteria:

* a score >5 on the PHQ-9 OR a score >5 on the GAD-7
* patient at Lurie Division of Adolescent and Young Adult Medicine
* provider agreement that this would be an appropriate intervention
* age between 13 and 25
* comfort speaking and reading in either English or Spanish

Exclusion Criteria:

* inability to speak and understand English or Spanish
* imminent risk for suicide as indicated by a "Yes" response to questions #5 on the Ask Suicide Questions (ASQ) Screener

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Short Mood and Feelings Questionnaire (SMFQ; Messer et al., 1995) | Pre-Intervention (baseline), immediately after the intervention, 12-week follow-up
  A 13-item questionnaire designed to assess depressive symptoms in youth. Total scores range from 0 to 26, with higher scores indicating greater depression severity (primary outcome).
Patient Health Questionnaire-9 (PHQ-9) | Pre-Intervention (baseline), 12-week follow-up
  A 9 item questionnaire that objectifies and assesses degree of depression severity. Total scores range from 0 to 27, with higher scores indicating greater depression severity.
Generalized Anxiety Disorder -7 (GAD-7) | Pre-Intervention (baseline), 12-week follow-up
  A 7 item questionnaire that measures severity of anxiety, mainly in outpatients. Total scores range from 0 to 21, with higher scores indicating greater anxiety severity.

SECONDARY OUTCOMES:
Dietary Restriction Screener - 2 (DRS 2) | Pre-Intervention (baseline), immediately after the intervention, 12-week follow-up
  This is a a single-item screener designed to identify individuals recently engaging in problematic restriction. The single item is "Have there been any times within the past month when you have eaten in this manner because you were concerned about your body shape and/or weight?" and has participants respond with a yes or a no.
Adult State Hope Scale | Pre-Intervention (baseline), immediately after the intervention, 12-week follow-up
  The 3-item State Hope Scale is a a dispositional self-report measure of agency. This scale can range from 3 to 24, with higher scores indicating higher levels of agency thinking.
Self-Hate Scale | Pre-Intervention (baseline), immediately after the intervention, 12-week follow-up
  The 7-item Self-Hate Scale is a brief, psychometrically valid measure of self-hate. Total scores are calculated as the mean of all items and scores are coded such that higher ratings indicate higher levels of self-hate (range 1-7).
Beck Hopelessness -4 | Pre-Intervention (baseline), immediately after the intervention, 12-week follow-up
  This four-item scale measures major aspects of hopelessness using true/false questions examining the respondent's attitude for the past week. This scale ranges from 0-4 such that higher scores reflect higher levels of hopelessness.
Program Feedback Scale | Immediately after the intervention
  The program feedback scale asks participants to rate agreement with seven statements indicating perceived acceptability and feasibility of their selected SSI (eg, "I enjoyed the program") on a 5-point Likert scale (1="really disagree"; 5="totally agree"). Means and standard deviations are calculated for each item (range 0-7), with a mean of 3.5 for each item indicating acceptability and feasibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Perczel Forintos D, Rozsa S, Pilling J, Kopp M. Proposal for a short version of the Beck Hopelessness Scale based on a national representative survey in Hungary. Community Ment Health J. 2013 Dec;49(6):822-30. doi: 10.1007/s10597-013-9619-1. Epub 2013 Jun 12. PMID 23756722
- [Background] Schleider JL, Mullarkey MC, Weisz JR. Virtual Reality and Web-Based Growth Mindset Interventions for Adolescent Depression: Protocol for a Three-Arm Randomized Trial. JMIR Res Protoc. 2019 Jul 9;8(7):e13368. doi: 10.2196/13368. PMID 31290406
- [Background] Schleider J, Weisz J. A single-session growth mindset intervention for adolescent anxiety and depression: 9-month outcomes of a randomized trial. J Child Psychol Psychiatry. 2018 Feb;59(2):160-170. doi: 10.1111/jcpp.12811. Epub 2017 Sep 18. PMID 28921523
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Haynos AF, Fruzzetti AE. Initial evaluation of a single-item screener to assess problematic dietary restriction. Eat Weight Disord. 2015 Sep;20(3):405-13. doi: 10.1007/s40519-014-0161-0. Epub 2014 Nov 21. PMID 25412874
- [Background] Beard C, Hsu KJ, Rifkin LS, Busch AB, Bjorgvinsson T. Validation of the PHQ-9 in a psychiatric sample. J Affect Disord. 2016 Mar 15;193:267-73. doi: 10.1016/j.jad.2015.12.075. Epub 2015 Dec 31. PMID 26774513
- [Background] Snyder CR, Sympson SC, Ybasco FC, Borders TF, Babyak MA, Higgins RL. Development and validation of the State Hope Scale. J Pers Soc Psychol. 1996 Feb;70(2):321-35. doi: 10.1037//0022-3514.70.2.321. PMID 8636885
- [Background] Eyre O, Bevan Jones R, Agha SS, Wootton RE, Thapar AK, Stergiakouli E, Langley K, Collishaw S, Thapar A, Riglin L. Validation of the short Mood and Feelings Questionnaire in young adulthood. J Affect Disord. 2021 Nov 1;294:883-888. doi: 10.1016/j.jad.2021.07.090. Epub 2021 Jul 29. PMID 34375216